CLINICAL TRIAL: NCT04930263
Title: A Study of the Individualized Walking Exercise Program on Memory, Subjective Cognitive Complaint, and Brain-derived Neurotrophic Factor Among Postmenopausal Hypertensive Women
Brief Title: Walking Exercise on Memory, Subjective Cognitive Complaint, and Brain-derived Neurotrophic Factor for Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201808096RINA
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-06

CONDITIONS: Hypertension
Keywords: Walking exercise; Memory; Hypertension; Brain-derived neurotrophic factor; Subjective Cognitive Complaint; Women
MeSH Terms: conditions — Hypertension | interventions — Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: We conduct a single-blinded, randomized controlled study. Sixty-six participants are randomly assigned to the experimental group and the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Experimental): Behavioral: walking exercise
  1. The intervention was 24 weeks walking intervention program with moderate-intensity, 5 sessions a week for 30 minutes per section
  2. individualized education
  3. telephone and social media counselling
  4. booklet guidance
  Interventions: Behavioral: Aerobic exercise
- control group (Active Comparator): Given routine care and life health manual for the participants.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Aerobic exercise — The intervention was 24 weeks walking exercise program. Participants exercised frequency at 5 sessions a week for 30 minutes per section with moderate-intensity and wearable device assisted. Each session consisted of a 5 minutes warm-up, moderate-intensity walking exercises and 5 minutes cool-down. The program included individualized education, telephone and social media counselling, and booklet guidance
  Arms: Aerobic exercise
Behavioral: control group — control group received routine care and a manual on healthy living
  Arms: control group

SUMMARY:
The purpose of this study is to determine the effect of 6-month aerobic walking program on memory, subjective cognitive complaints, and brain-derived neurotrophic factor for older hypertensive women. Participants will be randomly assigned to the experimental group and the control group. The intervention group will last for 24 weeks. The outcome measurements included memory, subjective cognitive complaints, and brain-derived neurotrophic factor.

DETAILED DESCRIPTION:
The purpose of this study is to explore an aerobic walking program on memory, subjective cognitive complaints, and brain-derived neurotrophic factor. In quantitative study with experimental design, qualified subjects will be randomly assigned to experimental or control group. Experimental subjects will perform six-month aerobic walking program and control group receive routine care. The outcome measurements included memory, subjective cognitive complaints, and brain-derived neurotrophic factor. Data will be collected at baseline, the end of the six-month intervention. Data will be analyzed using Generalized Estimation Equation evaluate the effect of the intervention program.

ELIGIBILITY:
Inclusion Criteria:

1. aged 60-80 years old,
2. a diagnosed of hypertension ≥ 6 months
3. self-reporting the signs of memory or thinking skills problems

Exclusion Criteria:

1. probable cognitive impairment as assessed by Montreal Cognitive Assessment ( < 24 points),
2. significant conditions limiting walking ability (e.g. musculoskeletal problems, visual impairment, etc.),
3. already participating in 30 minutes or more of moderate-intensity exercise five times a week
4. a history of severe cardiovascular disease,
5. a history of neurologic or psychiatric disorder such as stroke, head injury dementia, Parkinson disease, and depression.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 66 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Chen Chou, Principal Investigator — Nursing
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of eighty women with hypertension were screened in the study. Ten women refused and four women did not have the time. Only 66 were enrolled
Groups:
- Aerobic Exercise: Behavioral: walking exercise
  1. The intervention was 24 weeks walking intervention program with moderate-intensity, 5 sessions a week for 30 minutes per section
  2. individualized education
  3. telephone and social media counselling
  4. booklet guidance
  Aerobic exercise: The intervention was 24 weeks walking exercise program. Participants exercised frequency at 5 sessions a week for 30 minutes per section with moderate-intensity and wearable device assisted. Each session consisted of a 5 minutes warm-up, moderate-intensity walking exercises and 5 minutes cool-down.
Period: Overall Study
Arm/Group | Aerobic Exercise | Control Group
Started | 33 | 33
Completed | 30 | 28
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Control Group | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (6.5) | 69.8 (7.6) | 69.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 30 | 28 | 58
The Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment is a cognitive screening instrument created and validated. It is a 10-minute test of seven cognitive domains, including executive functions, naming, verbal memory registration and learning, attention, abstraction, 5-min delayed verbal memory, and orientation. The scores range from 0 to 30, higher score reflect to better global cognitive function.
  units on a scale | 26.8 (1.9) | 26.8 (1.8) | 26.8 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Memory Function
Description: The Hopkins Verbal Learning Test was administered to measure verbal learning and memory. The score is a sum of correct responses in each of three learning trial (encoding) (possible score 0 to 36 for summed recall of trials) and a delayed recall trial (possible score 0 to 12). Higher scores mean a better memory.
Time Frame: outcome measure at 24th week
Population: The Hopkins Verbal Learning Test , Post-test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise | Control Group
Number analyzed (Participants) | 30 | 28
score on a scale
  The Hopkins Verbal Learning Test total Recall | 25.5 (4.5) | 24.0 (4.5)
  The Hopkins Verbal Learning Test, delayed recall | 9.7 (2.4) | 9.0 (2.1)

2. Secondary Outcome: Brain-derived Neurotrophic Factor
Description: Blood sample will be collected. Plasma concentrate of Brain-derived neurotrophic factor will be analyzed by enzyme-linked immunosorbent assay
Time Frame: outcome measure at 24th week
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Aerobic Exercise | Control Group
Number analyzed (Participants) | 30 | 28
pg/ml | 206.0 (52.7) | 176.2 (72.2)

3. Secondary Outcome: Subjective Cognitive Complaints
Description: Cognitive Failures Questionnaire will be used to assess subjective cognitive impairment. Each item is rated from 0 to 4 with the total score calculated as the sum of all items ranging from 0 to 100 with higher scores indicating higher levels of cognitive failures.
Time Frame: outcome measure at 24th week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aerobic Exercise | Control Group
Number analyzed (Participants) | 30 | 28
score on a scale | 18.9 (11.2) | 20.5 (13.1)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Aerobic Exercise | Control Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT04930263/Prot_SAP_000.pdf